CLINICAL TRIAL: NCT05331573
Title: Parkinsonian Patients Treated With Apomorphine Pump: Observatory of Skin Lesions
Acronym: POLEMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/069/OB
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-03

CONDITIONS: Patients With Parkinson's Disease Treated With Apomorphine Pumps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: apomorphine pump — observationnal

SUMMARY:
Treatment with subcutaneous apomorphine will be initiated according to the usual procedures at each centre. Once the patient is included in the study, he/she will be followed for 24 months according to a schedule of visits corresponding to his/her follow-up care.

The procedures outside of the patient's usual care are only more in-depth clinical assessments and examinations (interviews with a nurse, skin lesion assessment scale, quality of life scales, neurological and cognitive assessment scales).

At each visit, the patient will be seen in consultation by a state-qualified nurse from the neurology department who will conduct

* nursing interviews to assess tolerance and compliance with treatment. She will also look for data concerning the flow rate, the duration of the subcutaneous apomorphine pump and the injection methods (material used, rotation of injection sites, massages).
* collection of adverse effects and changes in concomitant treatments.
* assessment of skin complications (number, location, characteristics: size, pain, inflammation).

For centres that do not have a nurse dedicated to monitoring these patients, the above procedure will be carried out by the neurologist.

In all cases, the patient will receive a consultation (in the department or remotely) by the neurologist.

The tests and scales performed at inclusion will be repeated at each six-monthly visit.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years,
* Diagnosis of Parkinson's disease according to the MDS criteria (2015),
* Patients with a prescription for subcutaneous apomorphine pump therapy,
* Patient having read and understood the information letter and having expressed oral non-opposition to the research.

Exclusion Criteria:

* Patient unable to express opposition or non-opposition,
* Patient not affiliated to the social security system,
* Pregnant woman or woman in labour or breastfeeding,
* Person deprived of liberty by an administrative or judicial decision,
* Person placed under court protection, guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease treated with apomorphine pumps
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
the occurrence of at least one painful | up to 24 weeks
  pain rating scale ≥ 1/10
the occurence of treatment discontinuation | up to 24 weeks
  skin nodule any size

SECONDARY OUTCOMES:
Assessment of nodules | at stopping apomorphine
  number, localisation
assessment of the pain of nodules or erythema | up to 24 weeks
  Visual Analogue Scale from 1 to 10:
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale | six-monthly visit
Hoehn and Yahr | six-monthly visit
Parkinson's Disease Questionnaire : quality of life scale, | six-monthly visit
Test of Montreal Cognitive Assessment | six-monthly visit

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Amien, Amiens
  - CHU Caen, Caen
  - CH de Dreux, Dreux
  - CHRU Lille, Lille
  - Hôpital St Vincent de Paul, Lille
  - Chu Rouen, Rouen
  - Clinique Saint Hilaire, Rouen

IPD SHARING:
Plan to Share IPD: No